CLINICAL TRIAL: NCT01979900
Title: Phase III Clinical Study of Efficacy and Safety of Mycobacterium Vaccae to Prevent Tuberculosis in High Risk Groups of Tuberculosis Infection
Brief Title: Phase III Clinical Study of Efficacy and Safety of Vaccae™ to Prevent Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government); Liuzhou Center for Disease Control and Prevention,China (Unknown); Rongshui County Disease Control and Prevention,China (Unknown); Liucheng County Disease Control and Prevention,China (Unknown); Jin Chengjiang Center for Disease Control and Prevention,China (Unknown); National Institutes for Food and Drug Control, China (Other); Air Force Military Medical University, China (Other); Simoon Record Pharma Information Consulting Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LTao
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2015-08

CONDITIONS: Tuberculosis
Keywords: TB Infection; Lesion Degree; Bacteriology Indicators; Cavity; Humoral Immunity; Cellular Immunologic Response
MeSH Terms: conditions — Tuberculosis | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccae (Experimental): Experiment group:One vial of Vaccae diluted with 1.0ml sterile water for injection, take deep coxal muscle injection after shaking well, once every 2 weeks, 6 times totally.
  Interventions: Drug: Vaccae
- Placebo (Placebo Comparator): Placebo group:One vial of placebo diluted with 1.0ml sterile water for injection, take deep coxal muscle injection after shaking well, once every 2 weeks, 6 times totally
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vaccae — One vial of Vaccae diluted with 1.0ml sterile water for injection, take deep coxal muscle injection after shaking well, once every 2 weeks, 6 times totally.
  Other Names: Mycobacterium vaccae for Injection
  Arms: Vaccae
Drug: placebo — One vial of placebo diluted with 1.0ml sterile water for injection, take deep coxal muscle injection after shaking well，once every 2 weeks, 6 times totally.
  Other Names: Vaccae Lyophilized stabilizers
  Arms: Placebo

SUMMARY:
Mycobacterium Vaccae for Injection (Trade Name "Vaccae") is a kind of bio-products developed by Anhui Zhifei Longcom Biopharmaceutical Co.,Ltd.,and got "The New Drug Certificate "in 1999. Vaccae has been approved for adjuvant therapy of tuberculosis(TB), and is also the only recommended drug in TB immunotherapy by WHO. It was approved for production and sale by Anhui Zhifei Longcom Biopharmaceutical Co.,Ltd. in 2001, and got favourable comment in therapy of tuberculosis.

The purpose of this study is to add new indications for Vaccae, mainly to prevent Tuberculosis for high risk groups of Tuberculosis Infection . In December 2012, China Food and Drug Administration approved of the plan "Phase III Clinical Study of Efficacy and Safety of Mycobacterium Vaccae to Prevent Tuberculosis in high risk groups of Tuberculosis Infection". In the test, 10,000 cases whose skin tests of PPD are strongly positive are enrolled. Using random, double-blind, and placebo-controlled methods, the study is carried out to evaluate the efficacy and safety of Vaccae in preventing Tuberculosis. Meanwhile, in this test, TB incidence and degree of pathological changes of experimental group are lower than that of control group, and no drug-related SAEs are reported in treatment groups.

DETAILED DESCRIPTION:
The Main Purpose of the Study:

- Evaluation of efficacy of Vaccae to prevent Tuberculosis in high risk groups of Tuberculosis Infection.

The Secondary Purpose of the Study:

* Evaluation of Lesion Degree ( Bacteriology Indicators, Cavity) of patients and its relationship with Skin Test results of TB-PPD after Injection of Vaccae into the high risk groups.
* Evaluation of Changes in Humoral Immunity and Cellular Immunologic Response Before and After Injection of Vaccae

Test Hypothesis:

In the test, TB incidence and degree of pathological changes of experimental group are lower than that of control group, and no drug-related SAEs are reported in treatment groups

Blinding and Random:

Using random, double-blind, and placebo-controlled methods, evaluation of the efficacy and safety of Vaccae.

Using block randomization method, a random sequence was generated by the statistics personnel in Fourth Military Medical University Clinical Evaluation Center using SAS9.1.3 statistical software

The Unblinding includes the first time of Unblinding and the second time of Unblinding. The first time of Unblinding only distinguish groups , and the second time of Unblinding will uncover the final Blind Codes.

The Blind Codes of the design produce at one time, and unblinding will be carried out respectively at the first year and the second year after the beginning of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 15 to 65 years old, all genders.
* Skin test of Tuberculin Pure Protein Derivative (TB-PPD) is strongly positive ( the average diameter of PPD skin test induration is greater than or equal to 15mm,and（or）local blisters, necrosis).
* Agreed to participate in the test and sign the informed consent.
* Subjects agreed to participate in the experiments and voluntarily signed the informed consent. (guardians of 15-17- year-old subjects should agree, meanwhile).
* The subjects should comply with the requirements of the clinical trial protocol and be Followed.
* Have not participated in any other clinical trial for nearly three months.
* Women of childbearing age from 15 to 49 years should agree with urine pregnancy tests and take effective birth control measures in two years after the medication.
* Axillary temperature is normal.

Exclusion Criteria:

The first injection drug exclusion criteria :

* Suffering from any other serious disease, e.g. during cancer treatment, autoimmune disease, progressive atherosclerosis, diabetes accompanied with complications, chronic obstructive pulmonary disease (COPD) needing oxygen therapy, acute or progressive liver or kidney disease, congestive heart failure, etc.
* Known allergy to experiment drugs
* People with history of specific diagnosis of TB, extrapulmonary tuberculosis or have been cured
* People have history of allergy, convulsions, epilepsy, cerebropathy, neurological symptoms and signs
* Patients who have impaired or abnormal immune function, e.g. patients treated with immunosuppressor or immunopotentiator, received immunoglobulin preparation or blood products or plasma extraction outside the gastrointestinal tract in 3 months, human immunodeficiency virus or related diseases
* Oral corticosteroids
* Patients who have been using oral corticosteroids for more than 1 week, or hormone medication in vitro for a long time
* Acute febrile illness and infection
* Pregnant or lactating women, or women who have birth plan in following 2 years
* Any other cases that may influence the test evaluation

The second-sixth injection drug exclusion criteria :

* Subjects whose compliance is poor, and can not take medicine on time or according to the amount
* Patients who are using medicine and food that can influence the result
* Pregnant subjects during the test
* Patients who are reluctant to continue and require exit

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2013-10; Primary Completion 2017-11-26 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
The whole TB incidence after injection of Vaccae | Terminal Stage: two years after the last group of subjects enrolled
  Medium-term: one year after the last group of subjects enrolled or after observation of 38 cases of the disease, Terminal Stage: two years after the last group of subjects enrolled or after observation of 76 cases of the disease

SECONDARY OUTCOMES:
Lesion degree (Bacteriology indicators, cavity) of patients | two years after the last group of subjects enrolled or after observation of 76 cases of the disease
  Medium-term: one year after the last group of subjects enrolled or after observation of 38 cases of the disease, Terminal Stage: two years after the last group of subjects enrolled or after observation of 76 cases of the disease
Systemic and local reactions and adverse events | within 30 days after last dosing
  within 30 days after last dosing
The relation between skin test results and paroxysm of TB-PPD | Terminal Stage: two years after the last group of subjects enrolled or after observation of 76 cases of the disease
  Medium-term: one year after the last group of subjects enrolled or after observation of 38 cases of the disease, Terminal Stage: two years after the last group of subjects enrolled or after observation of 76 cases of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Guoai Si, Director, Principal Investigator — Jin Chengjiang Center for Diseases Control and Prevention, Hechi, Guangxi; Mingqiang Li, Director, Principal Investigator — Jin Chengjiang Center for Diseases Control and Prevention, Liuzhou, Guangxi; Keshua Meng, Director, Principal Investigator — Rongshui County Diseases Control and Prevention, Liuzhou, Guangxi; Debiao Qiao, Director, Principal Investigator — Liucheng County Diseases Control and Prevention, Liuzhou, Guangxi
Locations (4):
- China (4):
  - Jin Chengjiang Center for Diseases Control and Prevention, Hechi, Guangxi, Hechi, Guangxi
  - Liucheng County Diseases Control and Prevention, Liuzhou, Guangxi, Liuchow, Guangxi
  - Liuzhou Center for Diseases Control and Prevention, Liuzhou, Guangxi, Liuchow, Guangxi
  - Rongshui County Diseases Control and Prevention, Liuzhou, Guangxi, Liuchow, Guangxi

REFERENCES:
- [Background] Moran-Mendoza O, Marion SA, Elwood K, Patrick DM, FitzGerald JM. Tuberculin skin test size and risk of tuberculosis development: a large population-based study in contacts. Int J Tuberc Lung Dis. 2007 Sep;11(9):1014-20. PMID 17705981
- See also: Center for drug evaluation, CFDA ,China — https://wbca.cde.org.cn/wbca/clinmain.do?method=edit&ckmIdCode=2A2F055FEFF749918149A70D4830FE3C